CLINICAL TRIAL: NCT03713307
Title: Macro and Micro Haemodynamic Responses to Shock in the Renal and Systemic Circulations; a Prospective Observational Study
Brief Title: Macro and Micro Haemodynamic Responses to Shock in the Renal and Systemic - MICROSHOCK - RENAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Royal Centre for Defence Medicine (Other Government)
Responsible Party: Sponsor
Other Study IDs: 246076
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-10

CONDITIONS: Acute Kidney Injury; Septic Shock
Keywords: Septic shock; acute kidney injury; haemodynamic monitoring; microcirculation
MeSH Terms: conditions — Acute Kidney Injury; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, plasma, serum, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational study of the state of the renal and systemic circulations in patients with early septic shock. Both macro and microvascular parameters will be assessed using echocardiography, sublingual incident dark field video-microscopy and renal contrast enhanced ultrasound. Patients will be categorised by KDIGO degree of kidney injury at Day 7 and stratified. Haemodynamic and perfusion based variables over time for these groups will be compared to assess the impact of changes in same on the development of AKI. Lab based work to quantify renal injury biomarkers will also be undertaken.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years Within 48 hours of ICU admission Evidence of suspected or confirmed infection Serial Organ Failure Assessment (SOFA) score increase of 2 or more (assuming baseline 0 if no previous measures) Requiring vasopressor therapy to maintain a MAP > 65mmHg Lactate > 2 mmol/l despite initial fluid resuscitation

Exclusion Criteria:

Known intolerance to Sonovue or any other ultrasound contrast agent Acute Respiratory Distress Syndrome Pregnancy Breast Feeding mothers Patients not expected to survive 24 h in whom the intent of treatment is palliative

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with early septic shock admitted to ICU
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
KDIGO AKI grade | Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watchorn J, Huang D, Bramham K, Hutchings S. Decreased renal cortical perfusion, independent of changes in renal blood flow and sublingual microcirculatory impairment, is associated with the severity of acute kidney injury in patients with septic shock. Crit Care. 2022 Sep 1;26(1):261. doi: 10.1186/s13054-022-04134-6. PMID 36050737